CLINICAL TRIAL: NCT05705908
Title: Effect of Foot Bath Using Warm Water and Lavender Essential Oil on Postoperative Sleep Quality and Pain: A Randomized Controlled Study
Brief Title: Effect of Foot Bath on Postoperative Sleep Quality and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Acibadem University, Asisst. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ATADEK 2021-19/19
Record Dates: First submitted 2022-05-25; First posted 2023-01-31 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Nursing Caries; Pain, Postoperative; Sleep Deprivation
Keywords: Sleep quality; pain management; post-operative care; foot bath
MeSH Terms: conditions — Pain, Postoperative; Sleep Deprivation; Sleep Initiation and Maintenance Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group - No foot bath (No Intervention): * 24 hours after surgery - did not give foot bath to patients
  * Pain was evaluated with VAS scale. Post-operative 24th hour, 28th hour, 32nd hour, 36th hour, 40th hour, 44th hour, 48th hour, 52nd hour, 56th hour, 58th hour, 62nd Hour, 64th Hour., 68th Hour, 72nd Hour
  * Sleep Questionnaire was administered at 08:00-09:00 in the morning when the patient woke up; 24th hour, 48 th hour, 72 th hour.
- Experimental Group- Hot Foot Bath 1 (Experimental): * Post operative 24th hour - 48 th hour - 72 nd hour - gave patients hot foot bath
  * Patient was seated in an upright position.
  * FM 4020 Grundig brand footbath device was used for the Hot Foot Bath.
  * It was filled with 40 degrees water, 20 cm (4 lt. of water)
  * Soaked in hot water up to the ankles
  * The foot bath was continued for 20 minutes with the feet in the device.
  * After 20 minutes, the patient's feet were dried with a towel.
  * After the foot bath pain was evaluated with VAS scale. Post-operative 24th hour, 28th hour, 32nd hour, 36th hour, 40th hour, 44th hour, 48th hour, 52nd hour, 56th hour, 58th hour, 62nd Hour, 64th Hour., 68th Hour, 72nd Hour
  * Sleep Questionnaire was administered at 08:00-09:00 in the morning when the patient woke up; 24th hour, 48 th hour, 72 th hour.
  Interventions: Other: Hot Foot Bath 1
- Experimental Group- Hot Foot Bath 2 (Experimental): * Post operative 24th hour - 48 th hour - 72 nd hour - gave patients hot foot bath with Lavender Essential Oil
  * Patient was seated in an upright position.
  * FM 4020 Grundig brand footbath device was used for the Hot Foot Bath.
  * It was filled with 40 degrees water, 20 cm (4 lt. of water)
  * Soaked in hot water up to the ankles
  * The foot bath with Lavender Essential Oil was continued for 20 minutes with the feet in the device.
  * After 20 minutes, the patient's feet were dried with a towel.
  * After the foot bath with Lavender Essential Oil pain was evaluated with VAS scale. Post-operative 24th hour, 28th hour, 32nd hour, 36th hour, 40th hour, 44th hour, 48th hour, 52nd hour, 56th hour, 58th hour, 62nd Hour, 64th Hour., 68th Hour, 72nd Hour
  * Sleep Questionnaire was administered at 08:00-09:00 in the morning when the patient woke up; 24th hour, 48 th hour, 72 th hour.
  Interventions: Other: Hot Foot Bath 2

INTERVENTIONS:
Other: Hot Foot Bath 1 — * Hot foot bath device has a built-in heater (max. 44°C),
  * Hot foot bath device has anti-slip base, vibration and 2 rotating massage rollers, digital display/control panel and timer (20-60 minutes).
  * It is filled with water at 40 degrees so that it passes the ankle of the patient by 20 cm (4 liters of water).
  Arms: Experimental Group- Hot Foot Bath 1
Other: Hot Foot Bath 2 — * Hot foot bath device has a built-in heater (max. 44°C),
  * Hot foot bath device has anti-slip base, vibration and 2 rotating massage rollers, digital display/control panel and timer (20-60 minutes).
  * It is filled with water at 40 degrees so that it passes the ankle of the patient by 20 cm (4 liters of water).
  * 3 drops of lavender essential oil were dripped in the water
  Arms: Experimental Group- Hot Foot Bath 2

SUMMARY:
One of the most common problems in patients in the postoperative period is pain and the associated deterioration in sleep quality. Deterioration in sleep quality can cause pain to be perceived more severely. It is recommended to use non-pharmacological approaches as well as pharmacological interventions in the management of these problems. This study was planned to determine the effect of hot foot bath and lavender essential oil foot bath application on postoperative sleep quality and pain in patients undergoing abdominal surgery.

DETAILED DESCRIPTION:
It was planned as a randomized controlled trial. The population of the study consisted of patients who underwent abdominal surgery in the General Surgery Service of a private health group hospital in Istanbul. Patients who met the inclusion criteria constituted the sample.

"Visual Comparison Scale-VAS" and "Richard-Campbell Sleep Scale" were used during data collection.

Visual Comparison Scale-VAS: It is a scale that starts with no pain and ends with unbearable. The VAS scale consists of a 10 cm long line. At one end of the line, "no pain" signals what may be at the other end of the "unbearable pain." The patient is asked to point to a point that indicates the current level of pain.

Richard-Campbell Sleep Scale: This scale consists of 6 items that evaluate the depth of night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep and the noise level of the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. According to the scale, the score in the range of "0-25" indicates very bad sleep, and the score in the range of "76-100" indicates very good sleep.

Foot bath was started as of the 24th hour after the operation. During the 3 days they were hospitalized, they had a foot bath evening before going to sleep (experimental group). Routine service applications were performed in the control group. In order to ensure the comfort of the experimental and control group patients and to minimize their exposure to the external environment, the patient rooms were kept clean, at a suitable temperature (23-25 degrees) and quiet.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Electively planned robotic and laparoscopic abdominal (colorectal, hepatobiliary, gastric and esophageal surgery, bariatric surgery, peritoneal membrane cancer) surgical operations
* Surgeries performed under general anesthesia
* Patients who have been hospitalized for at least 3 days after surgery
* Patients without a detected sleep disorder (Patients with Insomnia Severity Index score between 0-7) will be included in the study.

Exclusion Criteria:

* Patients who constantly take a foot bath
* Emergency surgeries
* Those with literacy disabilities
* Those with physical and mental disabilities
* Patients with diabetes for more than 10 years
* Patients with diabetic foot, neuropathy, foot pressure sores or any skin disease on their feet
* Those with vascular diseases
* Those who are allergic to lavender
* Those with neurological diseases (dementia, alzheimer, etc.)
* Those who regularly use sleep and psychoactive drugs
* Those who use drugs that affect sleep during hospitalization (sedatives, etc.)
* Patients who were transferred to the post-operative revision or general intensive care unit will not be included in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Change between Post-operative Pain Score | Post-operative Change between Pain Score; 24th hour, 28th hour, 32nd hour, 36th hour, 40th hour, 44th hour, 48th hour, 52nd hour, 56th hour, 58th hour, 62nd Hour, 64th Hour, 68th Hour, 72nd Hour (data collection will be finished here)
  The Pain scale - VAS scale consists of a 10 cm long line. At one end of the line, "no pain" signals what may be at the other end of the "unbearable pain." The patient is asked to point to a point that indicates the current level of pain.
  The difference between pain scores over 3 days will be evaluated in hospital Patient's pain was evaluated with VAS - 14 times after surgery. Immediately after surgery means 0th hour.
  These times; post-operative 24th hour, 28th hour, 32nd hour, 36th hour, 40th hour, 44th hour, 48th hour, 52nd hour, 56th hour, 58th hour, 62nd Hour, 64th Hour., 68th Hour, 72nd Hour.
  It will be measured for the last time at 72 hours and data collection will be finished here

SECONDARY OUTCOMES:
Change between Sleep Scale Score | Post-operative change between sleep scale score; 24th Hour, 48th Hour, 72th Hour (data collection will be finished here)
  Richard-Campbell Sleep Scale: This scale consists of 6 items that evaluate the depth of night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep and the noise level of the environment. Each item is evaluated on a chart between 0 and 100 using the visual analog scale technique. According to the scale, the score in the range of "0-25" indicates very bad sleep, and the score in the range of "76-100" indicates very good sleep.
  Sleep Scale was administered at 08:00-09:00 in the morning (when the patient woke up) in hospital - 3 times. Immediately after surgery means 0th hour.
  These times; post-operative 24th Hour, 48th Hour, 72th Hour. It will be measured for the last time at 72 hours and data collection will be finished here

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Uslu, Asisst Prof, Study Chair — Acıbadem Mehmet Ali Aydınlar Üniversitesi
Locations (1):
- Yasemin Uslu, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armat MR, Mortazavi H, Akbari H, Ebrahimzadeh Z. The effect of footbath on the quality of sleep in older adults: A pilot study. Geriatr Nurs. 2021 Sep-Oct;42(5):1178-1183. doi: 10.1016/j.gerinurse.2021.07.008. Epub 2021 Aug 20. PMID 34419870
- [Result] Talebi Ghadicolaei H, Heydary Gorji MA, Bagheri B, Yazdani Charati J, Hadinejad Z. The Effect of Warm Footbath on the Quality of Sleep on Patients with Acute Coronary Syndrome in Cardiac Care Unit. J Caring Sci. 2019 Sep 1;8(3):137-142. doi: 10.15171/jcs.2019.020. eCollection 2019 Sep. PMID 31598506
- [Result] Seyyedrasooli A, Valizadeh L, Zamanzadeh V, Nasiri K, Kalantri H. The effect of footbath on sleep quality of the elderly: a blinded randomized clinical trial. J Caring Sci. 2013 Nov 30;2(4):305-11. doi: 10.5681/jcs.2013.036. eCollection 2013 Dec. PMID 25276739
- [Result] Effati-Daryani F, Mohammad-Alizadeh-Charandabi S, Mirghafourvand M, Taghizadeh M, Bekhradi R, Zarei S. Effect of Lavender cream with or without footbath on sleep quality and fatigue in pregnancy and postpartum: a randomized controlled trial. Women Health. 2018 Nov-Dec;58(10):1179-1191. doi: 10.1080/03630242.2017.1414101. Epub 2018 May 22. PMID 29787355
- [Result] Kim HJ, Lee Y, Sohng KY. The effects of footbath on sleep among the older adults in nursing home: A quasi-experimental study. Complement Ther Med. 2016 Jun;26:40-6. doi: 10.1016/j.ctim.2016.02.005. Epub 2016 Feb 15. PMID 27261980